CLINICAL TRIAL: NCT06417177
Title: Impact of Early Aging and Menopause on the Vascular Responses to Hypoxia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jacqueline K Limberg, PhD, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2100208
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Aging; Menopause; Hypoxia; Vasodilation
MeSH Terms: conditions — Hypoxia; Aneurysm | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hypoxia (Experimental): Participants will be exposed to hypoxia (low oxygen air) using a mask.
  Interventions: Drug: Placebo; Drug: Propranolol; Drug: Gemtesa
- Cold pressor test (Experimental): Participants will be exposed to the cold pressor test (ice water on the foot).
  Interventions: Drug: Placebo; Drug: Propranolol; Drug: Gemtesa
- Hypercapnia (Experimental): Participants will be exposed to hypercapnia (high carbon dioxide air) using a mask.
  Interventions: Drug: Placebo; Drug: Propranolol; Drug: Gemtesa

INTERVENTIONS:
Drug: Placebo — Participants will receive a placebo in pill form.
Drug: Propranolol — Participants will receive oral propranolol (1 mg/kg).
Drug: Gemtesa — Participants will receive oral gemtesa (75 mg).

SUMMARY:
The purpose of this study is to examine hypoxic vasodilation and the role of beta-adrenergic receptors in younger premenopausal, perimenopausal, and older postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Female assigned at birth
* Pre, peri- or post-menopausal
* Healthy weight (BMI ≥18 and ≤30 kg/m2)

Exclusion Criteria:

* Male (assigned at birth)
* Pregnancy, breastfeeding
* Use of hormone replacement therapies
* Hysterectomy
* Body mass index >30 kg/m2
* Diagnosed sleep apnea
* Current smoking/Nicotine/Drug use
* Nerve/neurologic disease
* Cardiovascular, hepatic, renal, respiratory disease
* Blood pressure ≥140/90 mmHg
* Diabetes, Polycystic ovarian syndrome
* Communication barriers
* Prescription medications
* Malignant cancer

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Forearm blood flow | Change from baseline to 5 minutes.
  Blood flow in the forearm measured with venous occlusion plethysmography.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No